CLINICAL TRIAL: NCT01142895
Title: Simulated Usability Trial of the T-Slim Ambulatory Insulin Infusion Pump
Brief Title: Validation Study of G4 User Interface
Acronym: G4
Status: Completed | Type: Observational
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Kathryn Rieger, Tandem Diabetes care, Inc.
Other Study IDs: TDC-G4
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this simulated useability study is to demonstrate the user interface and software design mitigate potential safety concerns.

DETAILED DESCRIPTION:
These are the detailed descriptive planned outcomes of this useability study.

* To demonstrate that human-interface design mitigations lead to effective, efficient, and safe use.
* Validate that foreseeable misuse does not lead to a safety hazard or patient injury.
* Validate the effectiveness and comprehension of critical warnings and alerts, including vibratory, auditory, and textual cues.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetes mellitus

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Novice adult pumpers, experienced adult pumpers, and non-pumper adults
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual)